CLINICAL TRIAL: NCT05345275
Title: Assessment of Postoperative Pain in Children With Computer Assisted Facial Expression Analysis
Brief Title: Assessment of Postoperative Pain in Children With Facial Expression Analysis
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Ayla Irem Aydin, Principal Investigator, PhD, RN, Uludag University
Other Study IDs: 517517517
Record Dates: First submitted 2022-03-24; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pain, Postoperative
Keywords: children; facial expression analysis; machine learning; pain assessment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pain assessments: In the study, primarily the pain assessment data of children were collected. In these pain assessments, assessments of the child, mother, nurse and an independent observer were taken. Simultaneously, a video recording of the child's facial expressions was made.
  Interventions: Other: The facial expressions analyzed

INTERVENTIONS:
Other: The facial expressions analyzed — The facial expressions associated with pain were analyzed by the researchers in the OpenFace program. The patient's pain scores were estimated in the Python program by combining the numerical outputs of facial expression analyses with machine learning algorithms.

SUMMARY:
The present study was conducted to evaluate the use of computer-aided facial expression analysis to assess postoperative pain in children. The study population consisted of patients in the age group of 7-18 years who underwent surgery at Bursa Uludağ University Faculty of Medicine Health Application and Research Hospital Pediatric Surgery Clinic between November 2019 and June 2021. The sample of the study consisted of total 83 children who agreed to participate in the study and who met the sample selection criteria. Data were collected by the researcher using the Wong Baker Faces (WBS) pain rating scale and Visual Analog Scale (VAS). Data were collected from the child, mother, nurse, and one external observer. Facial action units associated with pain were used for machine estimation. OpenFace was used to analyze the child's facial action units and Python was used for machine learning algorithms. Intraclass correlation coefficient, Kappa coefficient, and linear regression analysis were used for statistical analysis of the data. The pain score predicted by the machine and the pain score assessments of the child, mother, nurse, and observer were compared.

ELIGIBILITY:
Inclusion Criteria:

* The patient is awake and oriented after the surgery,
* The patient must be within the first 12 hours after the operation and not be discharged before the first 36 hours after the operation,
* The patient is between the ages of 7-18,
* It is the mother's staying with the patient as a companion.

Exclusion Criteria:

* Presence of any facial anomalies that may alter facial expression analysis,
* The patient has neurological and mental disorders,
* Having regular opiate use in the last 6 months,
* These are surgical procedures that require the patient to be in a prone position.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study sample consisted of 7-18 age group patients who underwent surgery in the pediatric surgery clinic of a university hospital.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the first observation on pain assessment of children by human | after surgery in the first 12 hours
  WBS scales were used for pain assessment of children, mothers, nurses, and observers.
the first observation on pain assessment of children by human | after surgery in the first 12 hours
  VAS scales were used for pain assessment of children, mothers, nurses, and observers.
the second observation on pain assessment of children by human | after surgery 24.-36. range hours
  VAS scales were used for pain assessment of children, mothers, nurses, and observers.
the second observation on pain assessment of children by human | after surgery 24.-36. range hours
  WBS scales were used for pain assessment of children, mothers, nurses, and observers.
child's facial expressions | up to the first 36 hours.
  Facial action units associated with pain were used from the camera recordings of the child's facial expressions.

SECONDARY OUTCOMES:
pain assessment of children by machine | up to the first 36 hours.
  machine-estimated pain severity score from facial expression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludağ University, Bursa, Turkey (Türkiye)